CLINICAL TRIAL: NCT04200079
Title: Kingston COPD Cohort
Brief Title: Kingston Chronic Obstructive Pulmonary Disease (COPD) Multidimensional Long Term Follow up Cohort
Acronym: KCOCO
Status: Recruiting | Type: Observational
Sponsor: Dr. Juan Pablo de Torres Tajes (Other)
Responsible Party: Sponsor-Investigator, Dr. Juan Pablo de Torres Tajes, Professor, Queen's University
Organization: Queen's University (Other)
Other Study IDs: 43105
Record Dates: First submitted 2019-12-12; First posted 2019-12-16 (Actual); Last update posted 2021-09-14 (Actual); Status verified 2021-09

CONDITIONS: COPD; Emphysema
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Emphysema

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- COPD: Long term (at least 10 years) multidimensional (clinical, laboratory, physiological and radiological) follow up of chronic Obstructive Pulmonary Disease patients.

SUMMARY:
Background: Chronic Obstructive Pulmonary (COPD) patients are the paradigm of the chronic complex patient. Their follow up can sometimes be difficult and challenging (1). There are patients with recurrent exacerbations that put an enormous burden on health care resources (2). They also have multiple comorbidities (3) that can sometimes make their management difficult. In an attempt to coordinate all these efforts KGH, HDH and Providence Care have numerous essential resources to take care of COPD patients like the nurse navigators, nurse practitioners and the pulmonary rehabilitation program. These programs provide an excellent support to the clinical activity of Respirologists and other health care providers.

Rationale: The main rationale for the development of the Kingston COPD cohort is to translate that highly demanding clinical activity in a teaching and research oriented activity that could be used by clinicians, medical students, residents and fellows. Having a guideline complained established protocol in COPD patients that are usually follow at KGH and HDH could help in not only in unified the way COPD patients are seeing (preserving the importance of the personalized approach) but most importantly established a multidimensional (clinical, physiological, radiological, laboratory) database. This could help know not only the results of our clinical activity but also have a long term (>5yrs) database for clinical research projects in collaboration with national and international research groups. Therefore this proposal is important because it will help translate our busy daily clinical work in a highly productive teaching and research activity.

DETAILED DESCRIPTION:
Aims: establish a long term multidimensional follow up of a large COPD cohort of COPD patients in Kingston, Ontario.

Specific Objectives: 1. established a simple and easy to apply follow up protocol in COPD patients. 2. Hire a research assistant 3. Set up the database.

Data source: Patients included in the present cohort will be those usually follow at the Respirology clinic at Hotel Dieu Hospital in Kingston Ontario.

Data elements: this will include clinical, laboratory, physiological and radiological data.

Clinical: baseline and yearly evaluation. The following information will be collected and registered: Age, gender, history of prematurity and low weight at birth, maternal smoking during pregnancy, history of infections or wheezing during infancy, pack year history: (age of smoking initiation, years smoking, packs per day, age of quitting if quit), active or former smokers, use of vaping or marihuana?, registration of Comorbidities using the Copd cOmorbidiTy indEx COTE index, use of medications: LABA, LAMA, dual, LABA/ICS, ICS, Roflumilast, Erithromycin, NAC, etc, use of O2 at home: lt/min and duration, CPAP and BiPAP and pressures, degree of dyspnea measure by the Medical Research Council scale, height, weight, Body Mass Index, Free Fat Mass Index determined by electrical bioimpedance, handgrip, abdominal and pelvic girth.

Laboratory: baseline and yearly The following information from the patient chart will be collected and registered: CBC (including differential specifically eosinophilia), CRP, baseline alfa 1 AT levels (only baseline), fibrinogen, basal ABG.

Physiological information: yearly evaluation The following information will be collected and registered: FEV1, FVC, FEV1/FVC, TLC, IC/TLC, RV/TLC, DLCO, KCO. MIP, MEP, 6MWD with and without O2 in those O2 Sat 90% or lower. In a sample of interest full Cardiopulmonary exercise test.

Radiological information: Yearly Low dose chest CT The following information will be registered from the final reports of the chest CT: Emphysema presence, type, extent and localization, PulmArt/Ao diameter ratio measurement, presence of bronchiectasis (type and localization), presence of air trapping, presence (type and localization) of interstitial changes, presence of coronary calcifications, presence of osteoporosis, presence of lung nodules---- Lung cancer.

Data storage and identification Data will be stored in an encrypted file behind a firewall in a KGH server. For research purpose patient's information will be anonimized by using a study ID number that will be linked to the CR number of every patient in a different encrypted file. There will be no personal identifiable information during the entire process of each of the proposed studies.

Statistical analysis plan The description of the characteristics of the participants will follow the following methodology: qualitative data will be described using relative frequencies. We will use the Kolmogorov-Smirnov test (K-S) to determine if a quantitative variable has a normal distribution. Quantitative data with a normal distribution will be expressed using the mean and the standard deviation (SD).

When comparison between groups is planned the following methodological plan will be applied: quantitative data with non-normal distribution will be described with the median and the interquartile range (IQR). Differences will be compared with chi square for qualitative data or student t test and Mann-Whitney U test for quantitative data according to each variable distribution.

ELIGIBILITY:
Inclusion Criteria:

1. Patients ages between 40-85 years old.
2. Smoking history of at least 10 pack year history
3. Active of former smokers
4. Diagnosis of COPD according to the GOLD definition (4): post bronchodilator spirometry FEV1/FVC ≤0.70, including those with other associated respiratory diseases like asthma, bronchiectasis, stable lung cancer or Interstitial Lung Disease.
5. Ability to perform all study procedures (complete pulmonary function tests, six minute walking test (6MWT) and chest computed tomography) and provide/sign informed consent.

Exclusion Criteria:

1. Patients not willing to sign the consent form
2. Patients with a life expectancy of less than 3 yrs.
3. Patients in palliative care.
4. Patients with chronic airway obstruction ie: FEV1/FVC≤0.70 of other etiology and without a smoking history of less than 10 packs year history.
5. Patients unable ort not able to perform the pulmonary function test, the 6MWT or the chest CT.

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: COPD patients usually followed at a Respirology clinic
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2020-01-14 (Actual); Primary Completion 2030-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Mortality | 10 years
  Patients that will die during the follow up period
Exacerbations | 10 years
  Number of COPD exacerbations per year

CONTACTS AND LOCATIONS:
Overall Officials: Juan P de Torres, MD, Principal Investigator — Queen's University
Locations (1):
- KHSC, Kingston, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
Only on specific request